CLINICAL TRIAL: NCT04725461
Title: Low Cost Prosthetic Socket for Lower Limb Amputees
Brief Title: Low Cost Socket for Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Laura Miller, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00207623
Record Dates: First submitted 2021-01-15; First posted 2021-01-26 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Amputation; Amputation; Traumatic, Limb; Amputation, Traumatic
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low cost lower limb socket testing (Experimental): Fabrication and testing of a low cost lower limb prosthetic socket and ensure this socket has appropriate suspension, comfort and f unction for a transtibial amputee.
  Interventions: Device: Low cost lower limb prosthetic socket

INTERVENTIONS:
Device: Low cost lower limb prosthetic socket — A pre-made 3D printed cylinder used as an outer shell is selected for each subject based on their measurements. The space between the residual limb and the outer shell will be filled with an expanding polyurethane foam (Foam IT 8, Smooth On Inc.) that conforms to the residual limb and bonds with the outer shell to form a strong and lightweight socket. The foam forms a smooth surface against the protective sheath; the socket is fully formed once the foam has hardened to the 3D printed cylinder.
  A prefabricated supracondylar suspension cuff made of Dacron or nylon, or a commercially available suspension sleeve may be will be applied to the prosthetic socket to aid in suspension. Commercially available components, including the International Committee of the Red Cross (ICRC) transtibial polypropylene component system will be attached to the bottom of the socket to allow the patient to ambulate in the prosthesis.

SUMMARY:
The purpose of this research is to test an investigational fabrication system for transtibial prostheses. This fabrication method will be tested for comfort and function to determine feasibility of use for amputees in developing countries.

To address the need for high quality and affordable prosthetic technology in developing countries, the investigators have developed a simplified socket fitting protocol using expandable rigid foam. The foam is formed by mixing small amounts of two liquid components, which typically expands to several times its original volume.

DETAILED DESCRIPTION:
Millions of amputees in low-income nations lack access to prosthetic care. Conventional socket fabrication is complex, and the need for prosthetists is far greater than the throughput of existing clinician training programs. The first step in fitting a prosthetic limb is to fabricate the socket, which fits over the residual limb and acts as the interface between the residual limb and the prosthesis. The socket is the most custom component of the prosthetic system and must be comfortable to wear, easy to clean, and durable enough to withstand years of day-to-day use.

Simple and low-cost methods for socket fabrication and fitting would improve access to prosthetic care and could give many people in need their first opportunity to use a prosthesis. We have developed an easy-to-follow method that allows us to cast the limb in less than 30 minutes and finish the socket in 90 minutes, making it a practical choice for socket fitting in busy clinical settings, and where users are unable to return for multiple fittings. We have submitted a provisional US patent for our socket fabrication method.

We hypothesize that our novel method of fabrication for a low cost prosthesis can produce a device that has appropriate suspension, a comfortable interface, and requires little long term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputees having had their amputation at least 6 months prior, so that they have a relatively stable conical residual limb shape and can ambulate independently
* Currently has a well-fitting prosthesis- as defined by a self-reported Socket Comfort Score of at least a 6 out of 10
* K2, K3, K4 level ambulators
* Understands the English language

Exclusion Criteria:

* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate usable, reliable data. The ability to obtain relevant user feedback and informal discussion adds significant value to this study.
* Significant other comorbidity: Any other medical issues or injuries that would preclude completion of the study (e.g stroke, pacemaker placement, etc), or that would otherwise prevent acquisition of usable data by researchers.
* Bulbous residual limb shape causing inability to fit within system restrictions
* Open wounds on the residual limb
* Inability to understand the English language

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Socket Comfort Score with Experimental Low Cost Socket | Day 2
  The Socket Comfort Score will be used with the experimental low cost socket. This measure allows the subject to subjectively rate how comfortable they perceive their socket on a scale of 1 to 10, and will be administered pre and post physical outcome measures
Socket Comfort Score with Clinically Prescribed Socket | Day 2
  The Socket Comfort Score will be used with the subjects clinically prescribed prosthetic system. This measure allows the subject to subjectively rate how comfortable they perceive their socket on a scale of 1 to 10, and will be administered pre and post physical outcome measures

SECONDARY OUTCOMES:
Four Square Step Test | Day 2
  A clinical test of the ability to change directions while stepping.
L-Test of Functional Mobility | Day 2
  The L Test is a timed ambulation over 20 meters, which includes two sit to/from stand transfers and three turns.
2 Minute Walk Test | Day 2
  Individual walks without assistance for 2 minutes and the distance is measured.
Amputee Mobility Predictor | Day 2
  A questionnaire that measures the ambulatory potential of lower limb amputees. It requires the amputee to complete various tasks. Including sitting balance, reaching, transfers, sit to stand, and standing balance,

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States